CLINICAL TRIAL: NCT01089647
Title: Montelukast and Nasa ICS for Treatment of Mild Obstructive Sleep Apnea in Adults
Brief Title: Montelukast and Inhaled Nasal Steroid Tx in Adult Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romaker & Associates (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ann M. Romaker, MD, UMKC sleep fellowship program director, Romaker & Associates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Adult OSA drug study; IISP 37206 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Medical treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Budesonide; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- budesonide and montelukast (Active Comparator): treatment arm
  Interventions: Drug: budesonide and montelukast
- placebo (Placebo Comparator): sugar pill, salt water nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: budesonide and montelukast — budesonide aqua nasal spray 1 spray each nostril bid for 12 weeks Montelukast pill 10 mg po daily for 12 weeks
  Arms: budesonide and montelukast
Drug: Placebo — sugar pill po daily for 12 weeks salt water nasal spray 1 spray each nostril bid for 12 weeks
  Arms: placebo

SUMMARY:
In children with mild apnea combined therapy with an inhaled nasal steroid and a medication that decreased nasal congestion (montelukast) was shown to be effective. We are testing to see if this combination works in adults with mild apnea as well.

DETAILED DESCRIPTION:
40 adults with mild OSA (< 5 apneas/hypopneas per hour of sleep) will receive either a combination of two medicines that decrease nasal congestion-montelukast and nasal budesonide-or a placebo pill and nasal spray. After 3 months of therapy, a repeat sleep study will be done to determine the differences, if any, in the frequency of sleep disordered breathing in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 100 years
* RDI between 5 - 15
* all races
* both sexes

Exclusion Criteria:

* craniofacial, syndromic, neurological abnormalities
* current or previous use of Singular, Rhinocort within last 6 months
* acute upper respiratory infections
* recent nasal trauma, nasal surgery, nasal septum perforation
* known immunodeficiency or under going immunosuppressant therapy
* current therapy with drugs that interact with Montelukast or Budesonide

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Romaker, MD, Principal Investigator — Romaker & Associates
Locations (2):
- United States (2):
  - Romaker & Associates, Kansas City, Missouri
  - Romaker & Assoc, Kansas City, Missouri

REFERENCES:
- [Derived] Smith DF, Sarber KM, Spiceland CP, Ishman SL, Augelli DM, Romaker AM. Effects of Medical Therapy on Mild Obstructive Sleep Apnea in Adult Patients. J Clin Sleep Med. 2019 Jul 15;15(7):979-983. doi: 10.5664/jcsm.7876. PMID 31383235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four consecutive patients were recruited from the sleep medicine clinic at St. Luke's Health System from 24 June 2010 to 20 March 2013
Period: Overall Study
Arm/Group | Budesonide and Montelukast | Placebo
Started | 17 | 17
Completed | 13 | 13
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Budesonide and Montelukast | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 10 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 7 | 13 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 14 | 30
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease in the Number of Apnea and/or Hypopnea Events to <5 Per Hour of Sleep
Description: by decreasing nasal congestion, we hope to decrease the number of respiratory events per hour of sleep back to the normal range
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide and Montelukast | Placebo
Number analyzed (Participants) | 13 | 13
Participants | 5 | 3
Statistical Analysis 1: Comparison: Budesonide and Montelukast vs Placebo; Between-group comparisons at follow-up were made using a stepwise multivariable logistic model; Test type: Other; p = 0.946, ANOVA

ADVERSE EVENTS:
Arm/Group | Budesonide and Montelukast | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 2/13 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide and Montelukast (N=13) | Placebo (N=13)
nosebleed (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — epistaxis
lower leg swelling (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No